CLINICAL TRIAL: NCT01400698
Title: An Open Study of the Safety and Efficacy of Saizen®, (Recombinant Human Growth Hormone, r-hGH), in Children Born With Serious Intra-uterine Growth Retardation (IUGR) Treated to Final Height
Brief Title: Saizen in Intra-uterine Growth Retardation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20184
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Children Born With Serious Intra-uterine Growth Retardation
Keywords: Intra-uterine growth retardation (IUGR); Saizen; Recombinant human growth hormone (r-hGH); Final height; Bone age; SGA (Small for Gestational Age)
MeSH Terms: interventions — Human Growth Hormone

ARMS (3):
- Saizen® (Continuous or intermittent treatment) (Experimental)
  Interventions: Drug: Saizen® A
- Saizen® (Observed and then continuous or no treatment) (Experimental)
  Interventions: Drug: Saizen® B
- Observation only (Other)
  Interventions: Other: Observation only

INTERVENTIONS:
Drug: Saizen® A — Continuous or intermittent treatment with recombinant human Growth Hormone (r-hGH) 0.067 milligram/kilogram/day (mg/kg/day) subcutaneously (sc).
  Other Names: r-hGH; Somatropin
  Arms: Saizen® (Continuous or intermittent treatment)
Drug: Saizen® B — Observed until the first signs of puberty and then continuous treatment with r-hGH 0.067 mg/kg/day sc or observed without treatment.
  Other Names: r-hGH; Somatropin
  Arms: Saizen® (Observed and then continuous or no treatment)
Other: Observation only — Subjects were only observed.
  Arms: Observation only

SUMMARY:
Study of safety of Saizen® in children born with serious intra-uterine growth retardation (IUGR) treated to final height. An open, phase III study involving 17 centers in France.

The study enrolled children who have completed 3 or 2 years of treatment and at least one year of post treatment observation in the Sponsor Studies GF 4001 (Safety and Efficacy of Saizen in the Treatment of Young Children Born with Severe IUGR) or GF 6283 (Effect of Intermittent versus Continuous Saizen Therapy in Young Children Born with Severe IUGR), respectively.

Detailed description: Serious IUGR is a syndrome characterized by low birth length and weight for gestational age (less than 10 percentile). The secretion of growth hormone in response to provocative stimuli (e.g. arginine, insulin) is normal in these children. Apart from low birth weight, children born with IUGR may have minor or major malformations.

A catch-up period with a supraphysiological growth velocity generally occurs during the first 6 to 24 months of life in 80 to 90 percent (%) of these children. This generally allows them to reach normal height. That means that conversely, approximately 10 to 20% of children do maintain a statural handicap. Puberty occurs at a normal age and the retardation in bone maturation present during the first years of life disappears very quickly. This leads to short adult stature in subjects who have not shown spontaneous catch-up during the first years of life. A safe and effective means of promoting growth without accelerating the timing or tempo of puberty would therefore be desirable.

ELIGIBILITY:
Inclusion Criteria:

* Previous inclusion, good compliance and normal completion of GF4001 or GF6283 in the treatment of growth failure in children born with serious IUGR (3-year continuous r-hGH treatment in GF4001 or 2-year continuous or intermittent r-hGH treatment in GF6283).
* Increase in height greater than 0.5 standard deviation (SD) during the first 2 years of r-hGH treatment in GF4001 or after 2 years of continuous or intermittent r-hGH treatment in GF6283.
* A written Informed Consent at the beginning of the pre-study visit must be obtained from the parent(s)/legal guardian(s), with the understanding that consent may be withdrawn by the subject or parents at any time without prejudice to their future medical care. Children able to understand the trial should personally sign and date the written informed consent, too.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known multiple malformation syndrome with severe psychomotor retardation and/or body hemihypertrophy.
* Severe psychomotor retardation.
* Severe congenital malformations.
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 1998-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Serono S.A., Geneva

REFERENCES:
- [Background] Sempé M, Pédron G, Roy-Pernot M-P. Auxologie, méthode et séquences. Paris: Theraplix, 1979.
- [Result] Simon D, Leger J, Fjellestad-Paulsen A, Crabbe R, Czernichow P; SGA Study Group. Intermittent recombinant growth hormone treatment in short children born small for gestational age: four-year results of a randomized trial of two different treatment regimens. Horm Res. 2006;66(3):118-23. doi: 10.1159/000093832. Epub 2006 Jun 12. PMID 16772718
- [Result] Fjellestad-Paulsen A, Czernichow P, Brauner R, Bost M, Colle M, Lebouc JY, Lecornu M, Leheup B, Limal JM, Raux MC, Toublanc JE, Rappaport R. Three-year data from a comparative study with recombinant human growth hormone in the treatment of short stature in young children with intrauterine growth retardation. Acta Paediatr. 1998 May;87(5):511-7. doi: 10.1080/08035259850158209. PMID 9641731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed 3 or 2 years treatment and at least 1 year post treatment observation in Sponsor Studies GF 4001 (Safety and Efficacy of Saizen in the Treatment of Young Children Born with Severe IUGR) or GF 6283 (Effect of Intermittent versus Continuous Saizen Therapy in Young Children Born with Severe IUGR), respectively were enrolled.
Groups:
- Saizen® Continuous (A1): Participants with bone age less than or equal to (<=) 12 years for girls or 14 years for boys and height <=-2 standard deviation (SD) received continuous treatment with recombinant human Growth Hormone (r-hGH) 0.067 milligram/kilogram/day (mg/kg/day) subcutaneously (sc) until they reached final height for a maximum duration of 10.6 years.
- Saizen® Intermittent (A2): Participants with bone age <=12 years for girls or 14 years for boys and height <=-2 SD received intermittent treatment with r-hGH 0.067 mg/kg/day sc until they reached final height for a maximum duration of 10.6 years. Intermittent treatment was given on an individual basis depending on the height achieved during the study.
- Observed, Not Randomized (B0): Participants with bone age <=12 years for girls or 14 years for boys and height greater than (>) -2 SD were observed until first signs of puberty but not randomized.
- Observed Then Randomized to Saizen® (B1): Participants with bone age <=12 years for girls or 14 years for boys and height >-2 SD were observed until first signs of puberty and if remained at a height >-2 SD, were randomized to receive continuous treatment with r-hGH 0.067 mg/kg/day sc until they reached final height for a maximum duration of 10.6 years. Participants whose height fell to <=-2 SD before the first sign of puberty, were randomized to either Saizen® Continuous (A1) or Saizen® Intermittent (A2) treatment group.
- Observed Then Randomized to Observation (B2): Participants with bone age <=12 years for girls or 14 years for boys and height >-2 SD were observed until first signs of puberty and if remained at a height >-2 SD, were randomized to observation group with no treatment until they reached final height for a maximum duration of 10.6 years. Participants whose height fell to <=-2 SD before the first sign of puberty, were randomized to either Saizen® Continuous (A1) or Saizen® Intermittent (A2) treatment group.
- Observation (C): Participants with bone age >12 years for girls or 14 years for boys or refused to be treated in any of the above groups were followed without treatment until they reached final height for a maximum duration of 10.6 years.
Period: Overall Study
Arm/Group | Saizen® Continuous (A1) | Saizen® Intermittent (A2) | Observed, Not Randomized (B0) | Observed Then Randomized to Saizen® (B1) | Observed Then Randomized to Observation (B2) | Observation (C)
Started | 23 | 23 | 2 | 14 | 14 | 15
Completed | 8 | 12 | 0 | 6 | 7 | 9
Not Completed | 15 | 11 | 2 | 8 | 7 | 6
Not completed — Lost to Follow-up | 2 | 5 | 2 | 1 | 4 | 3
Not completed — Withdrawal by Subject | 8 | 2 | 0 | 4 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Non-compliance | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 4 | 2 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Final Height: Not Treated: Includes all participants who did not achieve the final height during the study period and did not receive r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
- Non-Final Height: Treated: Includes all participants who did not achieve the final height during the study period and received r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
- Final Height: Not Treated: Includes all participants who achieved the final height during the study period and did not receive r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
- Final Height: Treated: Includes all participants who achieved the final height during the study period and received r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
- Total: Total of all reporting groups
Arm/Group | Non-Final Height: Not Treated | Non-Final Height: Treated | Final Height: Not Treated | Final Height: Treated | Total
Number analyzed (Participants) | 10 | 13 | 22 | 46 | 91
Age Continuous [Mean (Standard Deviation); unit: years] | 10.6 (3.0) | 9.2 (2.4) | 12.5 (3.1) | 9.5 (2.6) | 10.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10 | 21 | 41
  Male | 5 | 8 | 12 | 25 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 0 | 0 | 2
  Black | 0 | 0 | 0 | 1 | 1
  White | 8 | 13 | 22 | 45 | 88
Original Study [Number; unit: participants]
  GF4001 | 6 | 6 | 18 | 22 | 52
  GF6283 | 4 | 7 | 4 | 24 | 39
Birth Height [Mean (Standard Deviation); unit: cm] | 41.8 (4.3) | 42.2 (3.5) | 44.8 (3.4) | 42.3 (3.5) | 42.8 (3.7)
Birth Weight [Mean (Standard Deviation); unit: g] | 1848 (601.2) | 2076.9 (520.9) | 2312 (451.1) | 2030.9 (573.4) | 2085.3 (551.8)
Length of Gestation [Mean (Standard Deviation); unit: weeks] | 37 (2.9) | 37.3 (2.6) | 38.9 (1.5) | 37.9 (2.8) | 37.9 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Final Height
Description: Final height was defined as the height reached 1 year after height velocity (HV) was less than 2 centimeter/year (cm/year). Height velocity was the change in height since the previous year's measurement. Height was measured with a wall-mounted stadiometer (or in supine position if the participant's age was less than 3 years) and the measurement was repeated thrice by the same observer. The mean of the values obtained in the repeated measurements was taken for the analysis.
Time Frame: One year after final height was attained up to 10.6 years
Population: Intention-to-treat (ITT) population included all participants enrolled in this study. Safety population was identical in this study.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Non-Final Height: Not Treated | Non-Final Height: Treated | Final Height: Not Treated | Final Height: Treated
Number analyzed (Participants) | 10 | 13 | 22 | 46
cm | 145.90 (16.08) | 150.06 (12.89) | 153.27 (8.71) | 155.59 (8.38)

2. Primary Outcome: Height Standard Deviation Score (HSDS)
Description: HSDS was calculated as height minus reference mean height divided by SD of the reference mean height, both given by the reference growth table (Sempe) for the corresponding chronological age at the height measurement. Greater HSDS indicate greater height. (Sempe M et al., 1979)
Time Frame: One year after final height was attained up to 10.6 years
Population: ITT population included all participants enrolled in this study. Safety population was identical in this study.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Non-Final Height: Not Treated | Non-Final Height: Treated | Final Height: Not Treated | Final Height: Treated
Number analyzed (Participants) | 10 | 13 | 22 | 46
standard deviation score | -1.45 (0.76) | -1.90 (1.73) | -2.33 (1.01) | -1.99 (0.88)

3. Secondary Outcome: Parental Adjusted Height Standard Deviation Score (PAHSDS)
Description: PAHSDS is the distance between the participant's current and target heights, expressed in units of SD of the height distribution of the reference population. Target height is a measure of the height which the participant could hypothetically reach based only on his parents' heights. Target height standard deviation score (THSDS) was calculated as target height minus mean adult height of the reference population divided by SD of the mean adult height of the reference population.
Time Frame: One year after final height was attained up to 10.6 years
Population: ITT population included all participants enrolled in this study. Safety population was identical in this study.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Non-Final Height: Not Treated | Non-Final Height: Treated | Final Height: Not Treated | Final Height: Treated
Number analyzed (Participants) | 10 | 13 | 22 | 46
standard deviation score | -0.82 (0.59) | -1.52 (1.92) | -1.64 (1.61) | -1.24 (1.39)

4. Post Hoc Outcome: Duration of Treatment
Time Frame: Up to 10.6 years
Population: ITT population included all participants enrolled in this study. Safety population was identical in this study. Here, 'N' (number of participants analyzed) signifies those participants who were treated and hence, were evaluated for this measure.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Non-Final Height: Treated | Final Height: Treated
Number analyzed (Participants) | 13 | 46
years | 4.09 (2.92) | 4.51 (2.20)

5. Post Hoc Outcome: Duration of Participation in the Study
Time Frame: Up to 10.6 years
Population: ITT population included all participants enrolled in this study. Safety population was identical in this study. Here, 'N' (number of participants analyzed) signifies those participants who were evaluated for this measure.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Non-Final Height: Not Treated | Non-Final Height: Treated | Final Height: Not Treated | Final Height: Treated
Number analyzed (Participants) | 9 | 13 | 22 | 46
years | 2.08 (2.27) | 5.29 (2.89) | 4.10 (2.87) | 7.02 (2.06)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 30 after end of study
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Groups:
- Not Treated: Included all participants who did not receive r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
- Treated: Included all participants who received r-hGH 0.067 mg/kg/day sc either continuously or intermittently.
Arm/Group | Not Treated | Treated
Serious Adverse Events (participants affected / at risk) | 1/32 | 13/59
Other Adverse Events (participants affected / at risk) | 16/32 | 52/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Treated (N=32) | Treated (N=59)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Congenital jaw malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1)
Ear tube removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Keratoconus (Eye disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Treated (N=32) | Treated (N=59)
Pharyngitis (Infections and infestations) | 5 (6) | 9 (14)
Bronchitis (Infections and infestations) | 3 (6) | 8 (11)
Gastroenteritis (Infections and infestations) | 3 (3) | 7 (8)
Nasopharyngitis (Infections and infestations) | 0 (0) | 6 (11)
Influenza (Infections and infestations) | 0 (0) | 6 (8)
Ear infection (Infections and infestations) | 2 (3) | 4 (4)
Rhinitis (Infections and infestations) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (8)
Acne (Skin and subcutaneous tissue disorders) | 1 (2) | 6 (7)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4)
Headache (Nervous system disorders) | 1 (2) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No